CLINICAL TRIAL: NCT01947283
Title: Effectiveness of DECIDE in Patient-Provider Communication, Therapeutic Alliance & Care Continuation
Acronym: PCORI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Margarita Alegria, PhD, Chief, Disparities Research Unit, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CD-12-11-4187
Record Dates: First submitted 2013-09-18; First posted 2013-09-20 (Estimated); Results first posted 2019-03-08 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2018-11

CONDITIONS: Mental Disorders
Keywords: Patient-Provider Relationship; Shared Decision Making; Therapeutic Alliance; Mental Health; Minority Health; Patient Activation; Communication
MeSH Terms: conditions — Mental Disorders; Psychological Well-Being; Patient Participation; Communication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Intervention Patients & Providers (Experimental): Participants in this arm are intervention patients who will receive the DECIDE-PA intervention.
  These patients receive care from Intervention providers, who will receive the DECIDE-PC intervention.
  For intervention patients, the DECIDE PA is designed to help patients identify concerns about their condition or treatment and generate questions for providers regarding these concerns. The DECIDE PA intervention consists of 3-4 brief training sessions for patients delivered by Care Managers.
  For intervention providers, the DECIDE PC is designed to help providers improve therapeutic alliance, patient-provider communication, continuance in care, and satisfaction with services for patients in order to improve shared decision making.
  Interventions: Behavioral: DECIDE-PA
- Intervention Patients, Control Providers (Experimental): Participants in this arm are intervention patients who will receive the DECIDE-PA intervention.
  These patients receive care from Control providers, who will not receive the DECIDE-PC intervention.
  For intervention patients, the DECIDE PA is designed to help patients identify concerns about their condition or treatment and generate questions for providers regarding these concerns. The DECIDE PA intervention consists of 3-4 brief training sessions for patients delivered by Care Managers.
  Interventions: Behavioral: DECIDE-PA
- Control Patients, Intervention Providers (No Intervention): Participants in this arm are control patients who will not receive the DECIDE-PA intervention.
  These patients receive care from Intervention providers, who will receive the DECIDE-PC intervention.
  Control patients will receive a pamphlet called "Managing Your Mental Health Care." For intervention providers, the DECIDE PC is designed to help providers improve therapeutic alliance, patient-provider communication, continuance in care, and satisfaction with services for patients in order to improve shared decision making.
- Control Patients & Providers (No Intervention): Participants in this arm are control patients who will not receive the DECIDE-PA intervention.
  These patients receive care from Control providers, who will not receive the DECIDE-PC intervention.
  Control patients will receive a pamphlet called "Managing Your Mental Health Care."
- Non-Randomized Controlled Trial Patients (No Intervention): Participants in this arm are patients who did not participate in the Randomized Controlled Trial. One to two patients will be recruited for each enrolled provider (Control and Intervention). One clinical session per patient will be audio recorded. These clinical recordings will be used to provide feedback only for Intervention providers during part 1 of the DECIDE-PC intervention.
- Control Providers (No Intervention): Participants in this arm are providers who were randomized to the Control group. Control providers will not receive the DECIDE-PC intervention.
- Intervention Providers (Experimental): Participants in this arm are providers who were randomized to the Intervention group. Intervention providers will receive the DECIDE-PC intervention. The DECIDE PC is designed to help providers improve therapeutic alliance, patient-provider communication, continuance in care, and satisfaction with services for patients in order to improve shared decision making.
  Interventions: Behavioral: DECIDE-PC

INTERVENTIONS:
Behavioral: DECIDE-PA — The DECIDE-PA intervention teaches patients strategies for asking questions and communicating more effectively with their behavioral health care provider in order to improve shared decision making.
  Arms: Intervention Patients & Providers; Intervention Patients, Control Providers
Behavioral: DECIDE-PC — The DECIDE-PC intervention trains providers in patient-centered communication techniques and encourages providers to be receptive to patients who take a more active role during the clinical encounter in order to improve shared decision making.
  Arms: Intervention Providers

SUMMARY:
The purpose of this study is to learn more about how patients and healthcare providers interact in order to improve shared decision making. The investigators plan to test an intervention with two separate educational components-one for patients and one for providers-designed to encourage patients to ask questions and increase their level of involvement in their own care, while simultaneously training providers to be more receptive to patients' questions and concerns. Patients in the intervention group will receive three short (30-45 minute) trainings focused on developing and asking questions and will be interviewed three times over the course of the intervention to see how it has affected the quality of their care. Providers receiving the intervention will participate in three separate trainings, including a 12-hour group workshop, an additional two hour training, and six hours of individual instruction, including personalized feedback based on three audio-recorded patient visits. Previous studies looking at patient engagement and involvement in decision-making have shown that increased engagement is linked with improved outcomes, but that providers are sometimes not prepared to develop a collaborative relationship with patients. The investigators think that training both patients and providers to work together and communicate more effectively will improve quality of care and increase patient satisfaction more than interventions that focus on only one side of the clinical encounter. One of the major goals in studying patient-provider communication is to improve shared decision-making and see how it contributes to racial and ethnic disparities in mental health care, since minority patients have been shown to be less involved in care and have been shown to be perceived and treated differently by providers.

DETAILED DESCRIPTION:
The Center for Multicultural Mental Health Research (CMMHR) at Cambridge Health Alliance has recently been selected for funding by the Patient Centered Outcomes Research Institute (PCORI) to address the importance of patient-provider communication, shared decision making, and therapeutic alliance. Our research team demonstrated that a psycho-educational intervention (DECIDE-PA) improves patient activation and self-management in behavioral health care. However, the investigators found that providers were unresponsive or reacted negatively to patients' activation. In response, the investigators propose to combine DECIDE-PA with provider coaching (DECIDE-PC) to increase providers' receptivity to patient activation, and improve Shared Decision Making (SDM). The investigators also focus on quality of care, responding to clinic administrators who require interventions that improve quality of behavioral health care (mental health and substance treatments).

Aims: 1) Test the effectiveness of DECIDE PA+PC compared to usual care in improving SDM and patient-perceived quality of behavioral health care; 2) Test whether patient-centered communication and therapeutic alliance mediate the effect of the DECIDE PA+PC intervention on SDM; 3) Explore whether ethnic/racial or language matching between patient and provider moderates the effect of DECIDE PA+PC on SDM and quality of behavioral health care.

Intervention: The DECIDE PA+PC intervention is designed to improve the quality of mental health care for adult behavioral health patients by engaging minority participants in asking questions about their treatment. The intervention is administered to patients and providers and is designed to improve patient activation, self-management, and therapeutic alliance.

For patients, the DECIDE PA is designed to help patients identify concerns about their condition or treatment and generate questions for providers regarding these concerns. The DECIDE PA intervention consists of 3-4 brief training sessions for patients delivered by Care Managers.

For providers, the DECIDE PC is designed to help providers improve therapeutic alliance, patient-provider communication, continuance in care, and satisfaction with services for patients in concordant and discordant ethnic/racial dyads. The DECIDE PC training for providers consists of 1.5 days of training which focuses on augmenting patient-centered communication and therapeutic alliance as a possible underlying pathway by which SDM can take place. The training also addresses 1) lack of perspective taking; 2) frequent attributional errors that providers make; and 3) decreased receptivity to patient participation and collaboration in decision making. The training includes provider coaching totaling 15-20 hours.

Methods: For Aim 1, implement a randomized controlled trial comparing DECIDE-PA+PC with usual care on Shard Decision Making (SDM) and perceived quality of care. Identify treatment effects using multi-level models that account for nesting of observations, patients, providers, and clinics. For Aim 2, identify underlying mechanisms of the effect of the DECIDE-PA+PC intervention on SDM. Mediation analysis techniques are used that allow for rigorous testing of causal pathways and statistical adjustment for spurious correlation is used in instances where mediators and SDM measurement are contemporaneous. For Aim 3, expand Aim 1 models to test whether DECIDE-PA+PC impacts SDM and perceived quality differentially by ethnic/racial concordant/discordant dyads.

Usual Care: Usual care across clinics is described by clinicians as answering their patients' questions during the clinical encounter. Clinicians report that on average they perceive their patients as having limited involvement in decision-making. No DECIDE training for patients or providers will be applied to the control condition while the control provider and control patient are participating in the study. Once the control provider and control patient complete their participation in the study, they will be offered the DECIDE trainings.

Participating Sites: The investigators plan to administer the intervention to patients and providers at four participating Cambridge Health Alliance clinics, along with Beth Israel Deaconess Medical Center, Boston Children's Hospital, South Cove Community Health Center, Edward M Kennedy Health Center (Great Brook Valley Health Center), and two community health centers through Harbor Health Services (Neponset Health Center and Geiger Gibson Community Health Center).

ELIGIBILITY:
Patient Inclusion Criteria:

-Patients ages 18-80 who are receiving mental health treatment at one of the collaborating clinics.

Patient Exclusion Criteria:

-Patients will be excluded if they screen with mania, psychosis, or suicidality to ensure their safety and minimize the stress of receiving the intervention. Patients over the age of 65 will be assessed with a cognitive functioning screening instrument and excluded if possible cognitive impairment is indicated.

Provider Inclusion Criteria:

-Providers will be permitted to participate in this study if they are regular, paid staff that provide behavioral health services at any of the participating clinics. No other criteria will be required.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 481 (Actual)
Dates: Start 2013-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Alegria, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (8):
- United States (8):
  - South Cove Community Health Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - South End Community Health Center, Boston, Massachusetts
  - Family Services of Greater Boston, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (Ambulatory Psychiatry Unit), Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (Latino Mental Health), Boston, Massachusetts
  - Cambridge Health Alliance (Windsor Clinic, Macht Building, Central Street, Malden Primary Care Mental Health), Cambridge, Massachusetts
  - Edward M Kennedy Health Center (Great Brook Valley Health Center), Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alegria M, Nakash O, Johnson K, Ault-Brutus A, Carson N, Fillbrunn M, Wang Y, Cheng A, Harris T, Polo A, Lincoln A, Freeman E, Bostdorf B, Rosenbaum M, Epelbaum C, LaRoche M, Okpokwasili-Johnson E, Carrasco M, Shrout PE. Effectiveness of the DECIDE Interventions on Shared Decision Making and Perceived Quality of Care in Behavioral Health With Multicultural Patients: A Randomized Clinical Trial. JAMA Psychiatry. 2018 Apr 1;75(4):325-335. doi: 10.1001/jamapsychiatry.2017.4585. PMID 29466533
- See also: Disparities Research Unit (DRU) website — http://www.massgeneral.org/disparitiesresearch/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in August 2014 and ended in September 2016. Participants were recruited at behavioral health community clinics and psychiatric outpatient clinics in Massachusetts. Participants were assessed for eligibility and then randomized into a study arm.
Pre-assignment Details: Patients were excluded due to ineligibility (positive screening for mania, psychosis, and/or active suicidal ideation) or treatment discontinuation. Providers were excluded due to a lack of patients enrolled in the study. Both patient and provider study participants were excluded if they withdrew before randomization into a study arm.
Groups:
- Non Randomized Controlled Trial Patients: Participants in this arm are patients who did not participate in the Randomized Controlled Trial. One to two patients will be recruited for each enrolled provider (Control and Intervention). One clinical session per patient will be audio recorded. These clinical recordings will be used to provide feedback only for Intervention providers during part 1 of the DECIDE-PC intervention.
Period: Overall Study
Arm/Group | Intervention Patients & Providers | Intervention Patients, Control Providers | Control Patients, Intervention Providers | Control Patients & Providers | Non Randomized Controlled Trial Patients | Control Providers | Intervention Providers
Started | 89 | 68 | 83 | 72 | 95 | 34 | 40
Baseline Assessment | 89 | 68 | 83 | 72 | 0 | 34 | 40
Follow-up Assessment | 64 | 51 | 65 | 59 | 0 | 27 | 36
Clinical Recording | 65 | 54 | 68 | 57 | 0 | 0 | 0
End-of-Intervention Assessment | 74 | 53 | 73 | 66 | 0 | 32 | 33
In Analysis | 89 | 68 | 83 | 72 | 95 | 30 | 38
Completed NRCT Baseline Assessment | 0 | 0 | 0 | 0 | 95 | 0 | 0
Completed | 60 | 45 | 62 | 55 | 95 | 27 | 32
Not Completed | 29 | 23 | 21 | 17 | 0 | 7 | 8
Not completed — Death | 1 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 4 | 6 | 5 | 5 | 0 | 2 | 5
Not completed — Withdrawal by Subject | 10 | 8 | 4 | 1 | 0 | 0 | 2
Not completed — No Clinical Recording | 12 | 6 | 8 | 10 | 0 | 0 | 0
Not completed — Non-coding Clinical Recording language | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Missing Follow-up Assessment | 2 | 2 | 3 | 0 | 0 | 2 | 0
Not completed — No patients were enrolled in study | 0 | 0 | 0 | 0 | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Population: All participants who were enrolled in the study after the baseline interview and whose data was analyzed.
Groups:
- Intervention Providers & Patients: Participants in this arm are intervention patients who will receive the DECIDE-PA intervention.
  These patients receive care from Intervention providers, who will receive the DECIDE-PC intervention.
  For intervention patients, the DECIDE PA is designed to help patients identify concerns about their condition or treatment and generate questions for providers regarding these concerns. The DECIDE PA intervention consists of 3-4 brief training sessions for patients delivered by Care Managers.
  For intervention providers, the DECIDE PC is designed to help providers improve therapeutic alliance, patient-provider communication, continuance in care, and satisfaction with services for patients in order to improve shared decision making.
- Total: Total of all reporting groups
Arm/Group | Intervention Providers & Patients | Intervention Patients, Control Providers | Control Patients, Intervention Providers | Control Patients & Providers | Non Randomized Controlled Trial Patients | Control Providers | Intervention Providers | Total
Number analyzed (Participants) | 89 | 68 | 83 | 72 | 95 | 34 | 40 | 481
Age, Customized [Count of Participants; unit: Participants] — All participants who were enrolled in the study after the baseline interview and whose data was analyzed.
  Participants
    <=18 years | 1 | 1 | 2 | 0 | 2 | 0 | 0 | 6
    Between 18 and 65 years | 83 | 60 | 75 | 65 | 88 | 31 | 38 | 440
    >=65 years | 5 | 7 | 6 | 7 | 5 | 2 | 2 | 34
    Missing | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants] — All participants who were enrolled in the study after the baseline interview and whose data was analyzed.
  Participants
    Female | 58 | 47 | 56 | 51 | 57 | 24 | 32 | 325
    Male | 31 | 21 | 27 | 21 | 38 | 10 | 8 | 156
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — All participants who were enrolled in the study after the baseline interview and whose data was analyzed.
  Participants
    Hispanic or Latino | 41 | 26 | 34 | 29 | 38 | 8 | 7 | 183
    Not Hispanic or Latino | 48 | 42 | 49 | 43 | 57 | 26 | 33 | 298
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — All participants who were enrolled in the study after the baseline interview and whose data was analyzed.
  Participants
    American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
    Asian | 7 | 5 | 9 | 5 | 7 | 5 | 6 | 44
    Native Hawaiian or Other Pacific Islander | 2 | 0 | 2 | 1 | 1 | 0 | 0 | 6
    Black or African American | 14 | 6 | 12 | 6 | 9 | 2 | 1 | 50
    White | 36 | 32 | 31 | 33 | 43 | 22 | 30 | 227
    More than one race | 2 | 15 | 0 | 6 | 3 | 2 | 2 | 30
    Unknown or Not Reported | 28 | 10 | 28 | 21 | 32 | 3 | 1 | 123
Region of Enrollment [Number; unit: participants] — All participants who were enrolled in the study after the baseline interview and whose data was analyzed.
  participants
    United States | 89 | 68 | 83 | 72 | 95 | 34 | 40 | 481
Shared Decision Making Questionnaire (SDM-Q-9 Patient Version) [Mean (Standard Deviation); unit: units on a scale] — Evaluates patient SDM from a patient-provider visit. The 9 items are rated on a 6-point Likert scale ranging from 0 (completely disagree) to 5 (completely agree). Final scores are sum of rating, which ranges between 0 and 45. Converted to 0 (lowest level) and 100 (highest level). Population: For patients, row populations differ because of missing assessments. Patient assessments were not asked from providers.
  units on a scale
    number analyzed (Participants) | 86 | 67 | 83 | 71 | 91 | 0 | 0 | 398
    (all) | 77.15 (20.31) | 76.31 (18.27) | 77.82 (17.54) | 74.24 (21.04) | 75.4 (23.57) |  |  | 76.23 (20.32)
Perceptions of Care Survey - Global Evaluation of Care Scale (PoC) [Mean (Standard Deviation); unit: units on a scale] — Assesses patient perceptions of care in psychiatric settings. Includes 3 items, final scores are scored externally, and range from 0 (lowest quality) to 100 (highest quality). Population: For patients, row populations differ because of missing assessments. Patient assessments were not asked from providers.
  units on a scale
    number analyzed (Participants) | 89 | 67 | 83 | 71 | 95 | 0 | 0 | 405
    (all) | 90.78 (10.44) | 88.29 (12.33) | 90.74 (9.90) | 88.32 (12.45) | 92.75 (8.74) |  |  | 90.39 (10.77)
Patient Shared Decision Making in Behavioral Health (SDM-BH) Patient Version [Mean (Standard Deviation); unit: units on a scale] — Evaluates patient SDM from a patient-provider visit in behavioral health. The 10 items were developed by a research team and are rated on a 6-point Likert scale ranging from 1 (completely disagree) to 6 (completely agree). Final scores are sum of rating, which ranges between 6 and 60. A high score indicates good communication and that decision making was shared between patient and provider, as perceived by the patient. Population: Differences in number of patients analyzed reflect missing observations. Measure was not assessed for Non-RCT patients and providers.
  units on a scale
    number analyzed (Participants) | 62 | 39 | 57 | 45 | 0 | 0 | 0 | 203
    (all) | 49.35 (8.91) | 46.23 (8.26) | 48.58 (7.00) | 47.76 (9.30) |  |  |  | 48.18 (8.39)
Provider Shared Decision Making in Behavioral Health (SDM-BH) Provider Version [Mean (Standard Deviation); unit: units on a scale] — Evaluates provider SDM from a patient-provider visit in behavioral health. The 10 items were developed by a research team and are rated on a 6-point Likert scale ranging from 1 (completely disagree) to 6 (completely agree). Final scores are sum of rating, which ranges between 6 and 60. A high score indicates good communication and that decision making was shared between patient and provider, as perceived by the provider. Population: Provider measure not assessed from patients. For providers, differences reflect missing observations.
  units on a scale
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 21 | 26 | 47
    (all) |  |  |  |  |  | 46.29 (4.91) | 46.85 (3.97) | 46.60 (4.37)

OUTCOME MEASURES:

1. Primary Outcome: Shared Decision Making (OPTION) Independent Blind Coder Assessment Scores
Description: 12 items designed to assess SDM quality in medical visit. Rated on 5 point Likert scales ranging from 0 (behavior not observed) -- 4 (clinician exhibited behavior to high standard). Final scores are the sum of the rating and range from 0-44. Final scores were transformed to a scale that ranges from 0 (lowest SDM) - 100 (highest SDM).
Time Frame: Follow-up assessment (2 months)
Population: All participants who enrolled in the study after the baseline interview and whose data was analyzed. Measure for "Control Providers" and "Intervention Providers" is the average across all of their RCT patients, irrespective of whether they were intervention or control patients. Differences from overall numbers are due to missing observations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Patients & Providers | Intervention Patients, Control Providers | Control Patients, Intervention Providers | Control Patients & Providers | Non Randomized Controlled Trial Patients | Control Providers | Intervention Providers
Number analyzed (Participants) | 65 | 54 | 68 | 57 | 93 | 28 | 36
units on a scale | 36.31 (11.77) | 29.78 (10.53) | 34.50 (14.96) | 30.37 (13.54) | 32.37 (12.96) | 30.09 (12.12) | 35.39 (13.48)

2. Primary Outcome: Shared Decision Making Questionnaire (SDM-Q-9 Patient Version)
Description: Evaluates patient SDM from a patient-provider visit based on their perception of nine steps deemed essential to SDM in a clinical encounter. Rated on a 6-point Likert scale ranging from 0 (completely disagree) to 5 (completely agree). Final scores are sum of rating, which ranges between 0 and 45. Converted to 0 (lowest level) and 100 (highest level).
Time Frame: End-of-intervention Assessment (5 months)
Population: All participants who enrolled in the study after the baseline interview and whose data was analyzed. SDM-Q-9 patient version was not administered to providers. Measure was not assessed for Non-RCT patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Patients & Providers | Intervention Patients, Control Providers | Control Patients, Intervention Providers | Control Patients & Providers | Non Randomized Controlled Trial Patients | Control Providers | Intervention Providers
Number analyzed (Participants) | 72 | 52 | 72 | 66 | 0 | 0 | 0
units on a scale | 81.10 (17.77) | 77.5 (17.86) | 75.85 (19.91) | 76.75 (20.52) |  |  |

3. Primary Outcome: Provider Shared Decision Making in Behavioral Health (SDM -BH) Provider Version
Description: The 10 items was developed by research team to evaluate provider SDM from a patient-provider visit in behavioral health. Items are rated on a 6-point Likert scale ranging from 1 (completely disagree) to 6 (completely agree). Final scores are sum of rating, which ranges between 6 and 60. A high score indicates good communication and that decision making was shared between patient and provider, as perceived by the provider.
Time Frame: Follow-up Assessment (2 months)
Population: All participants who were enrolled in the study after the baseline interview and whose data was analyzed. Each enrolled provider completed a follow-up assessment for each of their enrolled patients, following the audio recording of their clinical session.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention Providers, Control Patients: Participants in this arm are control patients who will not receive the DECIDE-PA intervention.
  These patients receive care from Intervention providers, who will receive the DECIDE-PC intervention.
  Control patients will receive a pamphlet called "Managing Your Mental Health Care." For intervention providers, the DECIDE PC is designed to help providers improve therapeutic alliance, patient-provider communication, continuance in care, and satisfaction with services for patients in order to improve shared decision making.
Arm/Group | Intervention Patients & Providers | Intervention Patients, Control Providers | Intervention Providers, Control Patients | Control Patients & Providers | Non Randomized Controlled Trial Patients | Control Providers | Intervention Providers
Number analyzed (Participants) | 46 | 30 | 49 | 39 | 0 | 0 | 0
units on a scale | 41.26 (6.57) | 40.10 (7.45) | 41.96 (5.53) | 38.41 (7.11) |  |  |

4. Primary Outcome: Shared Decision Making Questionnaire (SDM-Q-9 Provider Version)
Description: Evaluates provider SDM from a patient-provider visit based on their perception of nine steps deemed essential to SDM in a clinical encounter. Rated on a 6-point Likert scale ranging from 0 (completely disagree) to 5 (completely agree). Final scores are sum of rating, which ranges between 0 and 45. Converted to 0 (lowest level) and 100 (highest level).
Time Frame: Follow-up Assessment (2 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Patients & Providers | Intervention Patients, Control Providers | Control Patients, Intervention Providers | Control Patients & Providers | Non Randomized Controlled Trial Patients | Control Providers | Intervention Providers
Number analyzed (Participants) | 63 | 50 | 67 | 57 | 0 | 0 | 0
units on a scale | 69.03 (12.51) | 69.60 (14.30) | 69.85 (10.14) | 68.46 (16.97) |  |  |

5. Primary Outcome: Perceptions of Care Survey - Global Evaluation of Care Scale (PoC)
Description: Assesses patient perceptions of care in psychiatric settings. Includes 3 items, final scores are scored externally, and range from 0 (lowest quality) to 100 (highest quality).
Time Frame: End-of-intervention Assessment (5 months)
Population: All participants who were enrolled in the study after the baseline interview and whose data was analyzed. PoC was not administered to providers. Measure was not assessed for Non-RCT patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Patients & Providers | Intervention Patients, Control Providers | Control Patients, Intervention Providers | Control Patients & Providers | Non Randomized Controlled Trial Patients | Control Providers | Intervention Providers
Number analyzed (Participants) | 74 | 52 | 72 | 66 | 0 | 0 | 0
units on a scale | 94.60 (7.64) | 91.15 (9.48) | 90.50 (12.45) | 89.00 (13.06) |  |  |

6. Primary Outcome: Patient Shared Decision Making in Behavioral Health (SDM -BH)- Patient Version
Description: The 10 items was developed by research team to evaluate patient SDM from a patient-provider visit in behavioral health. Items are rated on a 6-point Likert scale ranging from 1 (completely disagree) to 6 (completely agree). Final scores are sum of rating, which ranges between 6 and 60. A high score indicates good communication and that decision making was shared between patient and provider, as perceived by the patient.
Time Frame: End-of-intervention Assessment (5 months)
Population: All participants who were enrolled in the study after the baseline interview and whose data was analyzed. SDM-BH patient version was not administered to providers. Measure was not assessed for Non-RCT patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Patients & Providers | Intervention Patients, Control Providers | Control Patients, Intervention Providers | Control Patients & Providers | Non Randomized Controlled Trial Patients | Control Providers | Intervention Providers
Number analyzed (Participants) | 65 | 44 | 68 | 58 | 0 | 0 | 0
units on a scale | 51.46 (6.63) | 47.14 (10.54) | 50.28 (7.85) | 48.67 (7.89) |  |  |

ADVERSE EVENTS:
Time Frame: Recruitment (0 months) to Completion of Study Participation (6 months)
Arm/Group | Intervention Patients & Providers | Intervention Patients, Control Providers | Control Patients, Intervention Providers | Control Patients & Providers | Non-Randomized Controlled Trial Patients | Control Providers | Intervention Providers
All-Cause Mortality (participants affected / at risk) | 1/89 | 1/68 | 1/83 | 0/72 | 0/95 | 0/34 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/68 | 0/83 | 0/72 | 0/95 | 0/34 | 0/40
Other Adverse Events (participants affected / at risk) | 0/89 | 0/68 | 0/83 | 0/72 | 0/95 | 0/34 | 0/40

LIMITATIONS AND CAVEATS:
Due to research assistants being blinded to study assignment, 18.5% of intervention arm patients completed their Time 2 assessments before the patient intervention. This impacted patients by chance and does not invalidate effectiveness assessment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No